CLINICAL TRIAL: NCT01594580
Title: A Novel Agent to Decrease Contamination of Hospital Scrubs
Brief Title: Contamination of Hospital Scrubs
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Maryland, Baltimore (Other)
Responsible Party: Principal Investigator, J. Kristie Johnson, Assistant Professor, University of Maryland, Baltimore
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Prevention
Other Study IDs: HP-00051506
Record Dates: First submitted 2012-05-07; First posted 2012-05-09 (Estimated); Last update posted 2023-07-21 (Actual); Status verified 2023-07

CONDITIONS: Bacterial Contamination

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Antimicrobial impregnated scrubs (Experimental): Those randomized to this arm of the study will wear scrubs impregnated with an antimicrobial.
  Interventions: Other: Antimicrobial impregnated scrubs
- Non-impregnated scrubs (Placebo Comparator): Those randomized to this arm of the study will wear scrubs not impregnated with an antimicrobial.
  Interventions: Other: Non-impregnated scrubs

INTERVENTIONS:
Other: Antimicrobial impregnated scrubs — Scrubs are impregnated with an antimicrobial product
  Arms: Antimicrobial impregnated scrubs
Other: Non-impregnated scrubs
  Arms: Non-impregnated scrubs

SUMMARY:
This study will test if nurses wearing scrubs treated with an antimicrobial agent while performing patient care will:

- Decrease the amount of bacterial contamination on scrubs at the end of a typical hospital shift during routine use after home laundering

This study will gather information by obtaining swabs from scrubs treated with an antimicrobial and from non-treated scrubs.

DETAILED DESCRIPTION:
The outcome of interest is the contamination of scrubs with Staphylococcus aureus, Enterococcus species or Gram-negative bacteria as determined by surface swabs of healthcare worker scrubs after a full 8-hour shift. The outcomes will be analyzed both individually and collectively.

Contamination will be defined as:

- A swab that is determined to be positive for any Staphylococcus aureus, Enterococcus species, or Gram-negative bacteria after a hospital shift.

ELIGIBILITY:
Inclusion Criteria:

* Nursing staff engaging in direct patient care
* Working in select/participating intensive care and intermediate care units
* Working at least 8 day shifts in one month (study period)

Exclusion Criteria:

* Pregnant
* Unable to provide consent
* Unable to follow study schedule

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 111 (Actual)
Dates: Start 2012-04; Primary Completion 2012-12 (Actual); Study Completion 2012-12 (Actual)

PRIMARY OUTCOMES:
Bacterial contamination of scrubs | Outcome will be assessed at the end of the hospital shift ( approx 8 hours)
  Contamination will be defined as:
  * A swab that is determined to be positive for any of Staphylococcus aureus, Enterococcus species, or Gram-negative bacteria after a hospital shift.

CONTACTS AND LOCATIONS:
Overall Officials: J Kristie Johnson, PhD, Principal Investigator — University of Maryland, Baltimore